CLINICAL TRIAL: NCT01392794
Title: Bioequivalence Study of YM060 Orally-disintegrating Tablet and Conventional Tablet - Ingestion Without Water
Brief Title: A Study to Compare Oral Absorption of YM060 Between Orally-disintegrating Tablet (Without Water) and Conventional Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 060-CL-208
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Healthy; Plasma Concentration of YM060
Keywords: YM060; ramosetron; orally-disintegrating tablet; OD tablet; bioequivalence
MeSH Terms: interventions — ramosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- orally-disintegrating (OD) tablet precedence group (Experimental)
  Interventions: Drug: YM060
- conventional tablet precedence group (Experimental)
  Interventions: Drug: YM060

INTERVENTIONS:
Drug: YM060 — oral, without water
  Other Names: ramosetron; Irribow

SUMMARY:
A study to compare time-course changes of plasma concentration of YM060 after intake of conventional tablet and orally-disintegrating tablet. Orally-disintegrating tablets will be administered without water.

ELIGIBILITY:
Inclusion Criteria:

* healthy assessed by the principal investigator or sub-investigators
* non-smoking or stop smoking at least 90 days before the study
* body weight: over 50.0kg and less than 80.0kg
* body mass index (BMI): over 17.6 and less than 26.4

Exclusion Criteria:

* participated in another clinical trial (including a post-marketing clinical study) within 120 days before the study
* donated 400mL of whole blood within 90 days, 200mL of whole blood within 30 days or blood components within 14 days before the study
* received any drugs within 7 days before the study or going to receive any drugs
* deviance from normal range in vital signs (blood pressure, pulse rate, and body temperature) or 12-lead ECG
* deviance from normal range in lab-tests
* history of drug allergy
* history or current diagnosis of stomach, small intestine or large intestine diseases
* history or current diagnosis of inflammatory bowel disease (Crohn's disease or colitis ulcerative)
* history or current diagnosis of colitis ischemic
* history or current diagnosis of hepatic diseases
* history or current diagnosis of cardiovascular diseases
* history or current diagnosis of respiratory diseases
* history or current diagnosis of malignant tumor
* received ramosetron tablet

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Area under the curve of YM060 plasma concentration -time curve | up to 24 hours after administration
Maximal concentration of YM060 plasma concentration | up to 24 hours after administration

SECONDARY OUTCOMES:
Safety assessed by the incidence of adverse events, vital signs, lab-tests and 12-lead ECG | up to 24 hours after administration

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Tokyo, Japan